CLINICAL TRIAL: NCT02281292
Title: A Randomized, Sham Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Activity of Intravitreal LKA651 in Patients With Diabetic Macular Edema
Brief Title: A Study of the Safety and Tolerability of Intravitreal LKA651 in Patients With Diabetic Macular Edema
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Management Decision
Sponsor: Alcon Research (Industry)
Collaborators: Novartis Institutes for BioMedical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LKA651X-2101
Record Dates: First submitted 2014-10-30; First posted 2014-11-03 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; Intravitreal; Retina; Ophthalmology; Lucentis; OCT
MeSH Terms: interventions — Ranibizumab; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- LKA651 (Part 1) (Experimental): LKA651 ophthalmic solution in 1 of 5 concentrations, administered as a single IVT injection in the study eye
  Interventions: Biological: LKA651 ophthalmic solution
- Sham injection (Part 1) (Placebo Comparator): Sham injection in the study eye
  Interventions: Biological: Sham injection
- LKA651 and Lucentis (Part 2) (Experimental): LKA651 ophthalmic solution in 1 of 3 concentrations, administered as a single IVT injection in the study eye, followed by ranibizumab ophthalmic solution, 0.5 mg injection in the same eye 30 minutes later
  Interventions: Biological: LKA651 ophthalmic solution; Biological: Ranibizumab ophthalmic solution
- Sham injection and Lucentis (Part 2) (Placebo Comparator): Sham injection in the study eye, followed by ranibizumab ophthalmic solution, 0.5 mg injection in the same eye 30 minutes later
  Interventions: Biological: Ranibizumab ophthalmic solution; Biological: Sham injection

INTERVENTIONS:
Biological: LKA651 ophthalmic solution
  Arms: LKA651 (Part 1); LKA651 and Lucentis (Part 2)
Biological: Ranibizumab ophthalmic solution
  Other Names: Lucentis®
  Arms: LKA651 and Lucentis (Part 2); Sham injection and Lucentis (Part 2)
Biological: Sham injection — Mock injection administered as an empty hub without needle
  Arms: Sham injection (Part 1); Sham injection and Lucentis (Part 2)

SUMMARY:
The purpose of this study is to evaluate the initial safety of intravitreal (IVT) LKA651 and potential for use alone or in combination with Ranibizumab ophthalmic solution (Lucentis®) for the treatment of Diabetic Macular Edema (DME) in patients with symptomatic disease.

DETAILED DESCRIPTION:
This first-in-human study will be conducted in 2 parts. Part 1 is an ascending dose design to assess the safety, tolerability, pharmacodynamics and pharmacokinetics of various single IVT doses of LKA651 in up to 48 subjects with diabetic macular edema. Subjects will be randomized to receive active or sham injections in a 3:1 ratio. A total of 6 cohorts (8 subjects per cohort) may be enrolled in Part 1. Each subject will participate in a screening/eligibility period (up to 60 days), a treatment period (single day), and an 84 day follow up period. A total of up to 11 visits will take place, all on an out-patient basis. An independent data monitoring committee (DMC) will be chartered to review cumulative safety data and approve each dose escalation and cohort progression in this first-in-human trial.

Part 2 is a double-masked design to assess the safety/tolerability, pharmacokinetics and pharmacodynamics of a single IVT dose of LKA651 when co-administered with Lucentis®. A total of up to 3 cohorts (8 subjects per cohort) may be enrolled in Part 2. Each subject will participate in a screening/eligibility period (up to 60 days), a treatment period (combination therapy, single day), and an 84 day follow up period. A total of up to 11 visits will take place, all on an out-patient basis. For the LKA651 vs sham injections, the unmasked ophthalmologist is not permitted to do any of the assessments except for the injection (and an inspection of the injection site immediately following). All other ocular assessments after randomization will be conducted by a second ophthalmologist masked to the type of injection (active or sham). The Lucentis injection (Part 2) is given open label to all patients following either the LKA651 or sham injection.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained.
* Type 1 or type 2 diabetes that is actively managed by a physician and hemoglobin A1C ≤ 12% at screening/eligibility.
* Negative pregnancy test results at screening/eligibility and pre-injection on treatment day.
* Diabetic macular edema (DME) with center involvement in at least one eye, including those with focal or diffuse DME.
* ETDRS letter score in the study eye of 55 letters or worse (approximate Snellen equivalent of 20/80). The non-study eye (fellow eye) should be ≥ 60 letters or better (approximate Snellen equivalent of 20/63) at Day 1 pre-dose.
* Safe to withhold treatment of the study eye with laser photocoagulation, intravitreal steroid injection, or intravitreal vascular endothelial growth factor (VEGF) inhibitor (Part 1) for the duration of the study.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Proliferative diabetic retinopathy in the study eye, with the exception of tufts of neovascularization less than 1 disc area with no vitreous hemorrhage.
* Any progressive disease of the retina (e.g. uveitis, rod-cone dystrophy) or optic nerve (e.g. glaucoma) other than diabetic retinopathy.
* Any active infection involving ocular adnexa including infectious conjunctivitis, keratitis, scleritis, endophthalmitis, as well as idiopathic or autoimmune-associated uveitis in either eye.
* Ocular disorders in the study eye that may confound interpretation of study results, including retinal vascular occlusion, retinal detachment, macular hole, or choroidal neovascularization of any cause (e.g., AMD, ocular histoplasmosis, or pathologic myopia).
* Cataract surgery in the study eye, Yttrium-Aluminum-Garnet (YAG) laser capsulotomy or any intraocular surgery within the past 6 months preceding Day 1.
* Use of systemic anticoagulant therapy during the study, e.g., warfarin, heparin, etc. The use of aspirin is not an exclusion.
* Use of other investigational drugs at the time of enrollment, or within 5 half-lives of enrollment, whichever is longer; or longer if required by local regulations.
* Pregnant or nursing (lactating) women.
* Women of child-bearing potential, unless using highly effective methods of contraception during dosing of study treatment.
* Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with a serious adverse event (SAE) that, in the opinion of the investigator, is related to the study drug | Up to Day 85
Number of subjects experiencing a non-serious adverse event | Up to Day 85

SECONDARY OUTCOMES:
The area under the serum concentration-time curve from time zero to the time of the last quantifiable concentration [mass x time / volume] (AUC(0-tlast)) | Up to Day 85
  Contingent upon observed serum concentration levels
The area under the serum concentration-time curve from time zero to time 't' where t is a defined time point after administration [mass x time / volume] (AUC (0-t)) | Up to Day 85
  Contingent upon observed serum concentration levels
The observed maximum serum concentration following drug administration [mass / volume] (Cmax) | Up to Day 85
  Contingent upon observed serum concentration levels
The time to reach the maximum serum concentration after drug administration [time] (Tmax) | Up to Day 85
  Contingent upon observed serum concentration levels
The dose normalized observed maximum serum concentration following drug administration [mass*dose / volume] (Cmax/D) | Up to Day 85
  Contingent upon observed serum concentration levels
The dose-normalized area under the serum concentration-time curve from time zero to the time of the last quantifiable concentration [mass*dose x time / volume] (AUC/D) | Up to Day 85
Central subfield thickness | Up to Day 85
  Contingent upon observed serum concentration levels

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Scientist, CSI, ID/Ophtha, Study Director — Alcon Research